CLINICAL TRIAL: NCT00460408
Title: European Epidemiologic COHORT Study: A Prospective Epidemiologic COHORT Study Of Ocular Safety In Patients Receiving Macugen Injections For Neovascular Age-Related Macular Degeneration (AMD) In Europe
Brief Title: Ocular Safety Of Patients Receiving Macugen For Neovascular Age Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5751019
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-11

CONDITIONS: Macular Degeneration
Keywords: Macular degeneration; Safety; Non-interventional; Non-randomized
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational study, no comparator: Observational study of patients with AMD treated with Macugen, no comparator
  Interventions: Drug: Macugen

INTERVENTIONS:
Drug: Macugen — Intravitreal injection of Macugen 0.3mg/90ul every 6 weeks.

SUMMARY:
The study will provide additional safety data for specific safety events in persons receiving intravitreal injections. The Committee for Medicinal Products for Human Use (CHMP) is interested in obtaining additional safety information when Macugen is used in real world settings by practitioners in Europe treating patients with neovascular (wet) age-related macular degeneration (AMD). The study will provide information about physician practice patterns and characteristics of patients treated with Macugen.

DETAILED DESCRIPTION:
No comparator Patients with age-related macular degeneration

ELIGIBILITY:
Inclusion Criteria:

* Neovascular AMD patients who are eligible for Macugen therapy based on the approved label

Exclusion Criteria:

* Active or suspected ocular or periocular infection. Known hypersensitivity to the active substance or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2006-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Charleroi
  - Pfizer Investigational Site, Ieper
  - Pfizer Investigational Site, Lier
  - Pfizer Investigational Site, Turnhout
- Pfizer Investigational Site, Limassol, Cyprus
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Sønderborg, Denmark
- France (6):
  - Pfizer Investigational Site, Argonay
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Le Golfe Juan
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Rennes
- Germany (8):
  - Pfizer Investigational Site, Augsburg
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Konstanz
  - Pfizer Investigational Site, Ludwigshafen
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Weilheim
- Greece (7):
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Nikaia, Piraeus
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Heraklion
  - Pfizer Investigational Site, Ioannina
  - Pfizer Investigational Site, Kavala
  - Pfizer Investigational Site, Thessaloniki
- Pfizer Investigational Site, Waterford, Ireland
- Italy (8):
  - Pfizer Investigational Site, Arona, NO
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Cagliari
  - Pfizer Investigational Site, Monza, MI
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Rieti
  - Pfizer Investigational Site, Siena
- Poland (3):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Slovakia (7):
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Ružomberok
  - Pfizer Investigational Site, Trenčín
  - Pfizer Investigational Site, Žilina
- Spain (7):
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Alcalá de Henares, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Valladolid, Valladolid
- Sweden (2):
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Västerås

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751019&StudyName=Ocular%20Safety%20Of%20Patients%20Receiving%20Macugen%20For%20Neovascular%20Age%20Related%20Macular%20Degeneration

RESULTS

PARTICIPANT FLOW:
Groups:
- Macugen: The use and dosage recommendations for Macugen (pegaptanib sodium) was in accordance with the summary of product characteristics. Participants could have received study drug in one eye or both eyes.
- Macugen and Avastin: The use and dosage recommendations for Macugen (pegaptanib sodium) was in accordance with the summary of product characteristics. Avastin (bevacizumab) for treatment of neovascular age-related macular degeneration (AMD) is an off-label use. Participants could have received study drug in one eye or both eyes.
- Macugen and Lucentis: The use and dosage recommendations for Macugen (pegaptanib sodium) and Lucentis (ranibizumab) was in accordance with the summary of product characteristics. Participants could have received study drug in one eye or both eyes.
- Macugen and Other AMD Drugs: The use and dosage recommendations for Macugen (pegaptanib sodium) and other approved AMD drugs were in accordance with the summary of product characteristics. Avastin (bevacizumab) for treatment of neovascular AMD is an off-label use. Participants could have received study drug in one eye or both eyes.
Period: Overall Study
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Started | 403 | 16 | 75 | 7
Completed | 336 | 13 | 69 | 7
Not Completed | 67 | 3 | 6 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 7 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 31 | 0 | 0 | 0
Not completed — Insufficient clinical response | 5 | 1 | 5 | 0
Not completed — Other | 12 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs | Total
Number analyzed (Participants) | 403 | 16 | 75 | 7 | 501
Age, Customized [Number; unit: participants]
  less than or equal to (≤) 50 years | 5 | 0 | 0 | 0 | 5
  51 to 64 years | 68 | 1 | 9 | 1 | 79
  65 to 74 years | 121 | 7 | 19 | 2 | 149
  greater than or equal to (≥) 75 years | 209 | 8 | 47 | 4 | 268
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 11 | 46 | 5 | 307
  Male | 158 | 5 | 29 | 2 | 194
Smoking status [Number; unit: participants] — Data missing for 1 participant in Macugen monotherapy reporting group.
  participants
    Never smoked | 265 | 12 | 45 | 5 | 327
    Current smoker | 34 | 1 | 8 | 0 | 43
    Exsmoker | 103 | 3 | 22 | 2 | 130

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pertinent Ocular Adverse Events (POAEs) Per Injection
Description: POAEs: primarily endophthalmitis, as well as increased intraocular pressure (IOP), vitreous hemorrhage, traumatic cataract, retinal detachment, and retinal tear. Incidence of POAEs per injection equals (=) number of specific POAEs divided by the total number of injections received.
Time Frame: Baseline up to 2 years
Population: Safety Population: participants who received at least 1 Macugen (pegaptanib sodium) injection; in addition to endophthalmitis, results for POAE categories presented if number of specific POAEs was ≥1 in at least 1 reporting group.
Measure: Number; unit: percent per injection
Units Other Than Participants: Injections
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Number analyzed (Participants) | 403 | 16 | 75 | 7
Number analyzed (Injections) | 2975 | 137 | 623 | 80
percent per injection
  Increased IOP | 1.34 | 2.19 | 0.48 | 2.50
  Vitreous hemorrhage | 0.10 | 0.73 | 0 | 0
  Traumatic cataract | 0.13 | 0 | 0 | 0
  Retinal detachment | 0.03 | 0 | 0 | 0
  Retinal tear | 0.03 | 0 | 0 | 0
  Endophthalmitis | 0 | 0 | 0 | 0

2. Secondary Outcome: Incidence of POAEs Per Injection Reported by Gender (Males)
Description: POAEs: primarily endophthalmitis, as well as increased IOP, vitreous hemorrhage, traumatic cataract, retinal detachment, and retinal tear. Incidence of POAEs per injection = number of specific POAEs divided by the total number of injections received.
Time Frame: Baseline up to 2 years
Population: Safety Population subset of male participants; in addition to endophthalmitis, results for POAE categories presented if number of specific POAEs was ≥1 in at least 1 reporting group.
Measure: Number; unit: percent per injection
Units Other Than Participants: Injections
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Number analyzed (Participants) | 158 | 5 | 29 | 2
Number analyzed (Injections) | 1195 | 43 | 238 | 26
percent per injection
  Increased IOP | 1.67 | 0 | 0 | 0
  Vitreous hemorrhage | 0.25 | 2.33 | 0 | 0
  Traumatic cataract | 0.08 | 0 | 0 | 0
  Retinal detachment | 0.08 | 0 | 0 | 0
  Retinal tear | 0.08 | 0 | 0 | 0
  Endophthalmitis | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of POAEs Per Injection Reported by Gender (Females)
Description: as for outcome 2
Time Frame: Baseline up to 2 years
Population: Safety Population subset of female participants; in addition to endophthalmitis, results for POAE categories presented if number of specific POAEs was ≥1 in at least 1 reporting group.
Measure: Number; unit: percent per injection
Units Other Than Participants: Injections
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Number analyzed (Participants) | 245 | 11 | 46 | 5
Number analyzed (Injections) | 1780 | 94 | 385 | 54
percent per injection
  Increased IOP | 1.12 | 3.19 | 0.78 | 3.70
  Traumatic cataract | 0.17 | 0 | 0 | 0
  Endophthalmitis | 0 | 0 | 0 | 0

4. Secondary Outcome: Incidence of POAEs Per Injection Reported by Age Group (≤ 50 Years)
Description: as for outcome 2
Time Frame: Baseline up to 2 years
Population: Safety Population subset of participants ≤50 years old
Measure: Number; unit: percent per injection
Units Other Than Participants: Injections
Arm/Group | Macugen
Number analyzed (Participants) | 403
Number analyzed (Injections) | 34
percent per injection
  Endophthalmitis | 0
  Vitreous hemorrhage | 0
  Traumatic cataract | 0
  Increased IOP | 0
  Retinal detachment | 0
  Retinal tear | 0

5. Secondary Outcome: Incidence of POAEs Per Injection Reported by Age Group (51 to 64 Years)
Description: as for outcome 2
Time Frame: Baseline up to 2 years
Population: Safety Population subset of participants 51 to 64 years of age; in addition to endophthalmitis, results for POAE categories presented if number of specific POAEs was ≥1 in at least 1 reporting group.
Measure: Number; unit: percent per injection
Units Other Than Participants: Injections
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Number analyzed (Participants) | 68 | 1 | 9 | 1
Number analyzed (Injections) | 554 | 10 | 101 | 15
percent per injection
  Increased IOP | 2.17 | 0 | 0 | 0
  Retinal tear | 0.18 | 0 | 0 | 0
  Endophthalmitis | 0 | 0 | 0 | 0

6. Secondary Outcome: Incidence of POAEs Per Injection Reported by Age Group (65 to 74 Years)
Description: as for outcome 2
Time Frame: Baseline up to 2 years
Population: Safety Population subset of participants 65 to 74 years of age; in addition to endophthalmitis, results for POAE categories presented if number of specific POAEs was ≥1 in at least 1 reporting group.
Measure: Number; unit: percent per injection
Units Other Than Participants: Injections
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Number analyzed (Participants) | 121 | 7 | 19 | 2
Number analyzed (Injections) | 933 | 65 | 144 | 27
percent per injection
  Increased IOP | 2.04 | 4.62 | 0 | 0
  Vitreous hemorrhage | 0.11 | 1.54 | 0 | 0
  Traumatic cataract | 0.21 | 0 | 0 | 0
  Retinal detachment | 0.11 | 0 | 0 | 0
  Endophthalmitis | 0 | 0 | 0 | 0

7. Secondary Outcome: Incidence of POAEs Per Injection Reported by Age Group (≥ 75 Years)
Description: as for outcome 2
Time Frame: Baseline up to 2 years
Population: Safety Population subset of participants ≥ 75 years of age; in addition to endophthalmitis, results for POAE categories presented if number of specific POAEs was ≥1 in at least 1 reporting group.
Measure: Number; unit: percent per injection
Units Other Than Participants: Injections
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Number analyzed (Participants) | 209 | 8 | 47 | 4
Number analyzed (Injections) | 1454 | 62 | 378 | 38
percent per injection
  Increased IOP | 0.62 | 0 | 0.79 | 5.26
  Vitreous hemorrhage | 0.14 | 0 | 0 | 0
  Traumatic cataract | 0.14 | 0 | 0 | 0
  Endophthalmitis | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Serious Hypersensitivity Reactions
Description: Hypersensitivity reactions include Hypersensitivity, Drug hypersensitivity, Anaphylactic shock, Anaphylactic reaction, Anaphylactoid shock, Angioedema Anaphylactoid reaction, Blepharitis allergic, Dermatitis contact, Dermatitis allergic, Toxic skin eruption, Toxic epidermal necrolysis, Drug eruption, Erythema, Erythema multiforme, Tongue oedema, Pharyngeal oedema, Laryngeal oedema, Latex allergy, Paraesthesia oral, Paraesthesia mucosal, Urticaria, Stevens-Johnson syndrome, Rash, Skin reaction, Acute generalised exanthematous pustulosis, Drug rash with eosinphilia and systemic symptoms.
Time Frame: Baseline up to 2 years
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Number analyzed (Participants) | 403 | 16 | 75 | 7
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Macugen | Macugen and Avastin | Macugen and Lucentis | Macugen and Other AMD Drugs
Serious Adverse Events (participants affected / at risk) | 21/403 | 0/16 | 2/75 | 0/7
Other Adverse Events (participants affected / at risk) | 65/403 | 4/16 | 14/75 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macugen (N=403) | Macugen and Avastin (N=16) | Macugen and Lucentis (N=75) | Macugen and Other AMD Drugs (N=7)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Vitreous fibrin (Eye disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macugen (N=403) | Macugen and Avastin (N=16) | Macugen and Lucentis (N=75) | Macugen and Other AMD Drugs (N=7)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 1 | 0
Blindness (Eye disorders) | 1 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 3 | 0 | 0 | 0
Choroidal neovascularisation (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 5 | 1 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 2 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 4 | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Meibomianitis (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Ocular hypertension (Eye disorders) | 5 | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 3 | 0 | 1 | 0
Scotoma (Eye disorders) | 0 | 0 | 1 | 0
Vitreous disorder (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 2 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 1 | 0
Injection site inflammation (General disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Ear infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Keratitis herpetic (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Intraocular pressure decreased (Investigations) | 1 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 26 | 2 | 2 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Convulsions local (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.